CLINICAL TRIAL: NCT03143751
Title: Continuous Hyperosomolar Therapy for Traumatic Brain-injured Patients Study Protocol for a Multicenter Randomized Open-label Trial With Blinded Adjudication of Primary Outcome
Brief Title: Continuous Hyperosomolar Therapy for Traumatic Brain-injured Patients
Acronym: COBI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC16_0474
Record Dates: First submitted 2017-04-28; First posted 2017-05-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Moderate to Severe Traumatic Brain Injury

STUDY DESIGN:
Who Masked: Participant
Masking Description: Masking: Open label , Masked Roles: Subject and Outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous hyperosmolar therapy (Experimental): Standard cares plus continuous hyperosmolar therapy (NaCl20%)
  Interventions: Drug: NaCl20% (Continuous hyperosmolar therapy)
- Control (No Intervention): Standard cares alone.

INTERVENTIONS:
Drug: NaCl20% (Continuous hyperosmolar therapy) — Early intravenous administration (<24 hours after traumatic brain injury) of NaCl20% for a minimal duration of 48 hours (continued for as long as is necessary to prevent intracranial hypertension)
  1-hour bolus (15 g if Na+ < 145 mmol/L; 7.5 g if 145 < Na+ < 150 mmol/L; or no bolus) followed by 1 g/hour as long as Na+< 150 mmol/L, reduced to 0.5 g/L if 150 < Na+ < 155 mmol/L, Discontinuation when 155 mmol/L<Na+
  Arms: Continuous hyperosmolar therapy

SUMMARY:
Traumatic brain injury (TBI) is a major cause of death and severe prolonged disability. Intracranial hypertension (ICH) is a critical risk factor of bad outcomes after TBI. Continuous infusion of hyperosmolar therapy has been proposed for the prevention or the treatment of ICH. Whether an early administration of continuous hyperosmolar therapy improves long term outcomes is uncertain. The aim of the current study is to assess the efficiency and the safety of continuous hyperosmolar therapy in TBI patients.

The COBI trial is the first randomized controlled trial powered to investigate whether continuous hyperosmolar therapy in TBI patients improve long term recovery.

Hypothesis

Patients treated with early continuous hyperosmolar therapy have reduced morbidity and mortality rates compared to those receiving standard care alone after traumatic brain injury.

Research Questions

1. Does early continuous hyperosmolar therapy reduce morbidity and mortality rates at 3 and 6 months after TBI assessed by the GOSE questionnaire?
2. Does early continuous hyperosmolar therapy prevent intracranial hypertension?

DETAILED DESCRIPTION:
Background Traumatic brain injury (TBI) is a major cause of death and severe prolonged disability. Intracranial hypertension (ICH) is a critical risk factor of bad outcomes after TBI.

Continuous infusion of hyperosmolar therapy has been proposed for the prevention or the treatment of ICH. Whether an early administration of continuous hyperosmolar therapy improves long term outcomes is uncertain. The aim of the current study is to assess the efficiency and the safety of continuous hyperosmolar therapy in TBI patients.

Methods The COBI (Continuous hyperosmolar therapy in traumatic brain-injured patients) trial is a multicenter, randomized, controlled, open-label, two-arms study with blinded adjudication of primary outcome. Three hundred and seventy patients hospitalized in Intensive Care Unit with a traumatic brain injury (Glasgow Coma Scale ≤ 12 and abnormal brain CT-scan) are randomized in the first 24 hours following trauma to standard care or continuous hyperosmolar therapy (NaCl 20%) plus standard care. Continuous hyperosmolar therapy is maintained for at least 48 hours in the treatment group and continued for as long as is necessary to prevent intracranial hypertension. The primary outcome is the score on the Extended Glasgow Outcome Scale (GOS-E) at 6 months. The treatment effect is estimated with ordinal logistic regression adjusted for pre-specified prognostic factors and expressed as a common odds ratio.

Discussion The COBI trial is the first randomized controlled trial powered to investigate whether continuous hyperosmolar therapy in TBI patients improve long term recovery.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Moderate to severe traumatic brain injury defined as the association of a Coma Glasgow Scale ≤ 12 together with a traumatic abnormal brain CT-scan
* Time to inclusion inferior to 24 hours
* Informed consent (or emergency procedure)

Exclusion Criteria:

* dependence for daily activity
* Coma Glasgow Scale of 3 and fixed dilated pupils
* associated cervical spine injury
* imminent death and do-not-resuscitate orders
* pregnancy.
* Major not legally responsible
* Oedemato-ascitic decompensation of hepatic cirrhosis
* State of hydro-sodium retention secondary to heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Score on the Extended Glasgow Outcome Scale (GOS-E) at 6 months | 6 months
  The GOS-E is a scale measuring the neurological recovery after traumatic brain injuries

SECONDARY OUTCOMES:
Mortality rate in ICU | 3 months
Mortality rate in ICU | 6 months
GOS-E | 3 months
  The GOS-E is a scale measuring the neurological recovery after traumatic brain injuries
functional independence measure : ADL (Activities of Daily Living) of Katz | 3 months
  Scale measuring the autonomy of patient
functional independence measure : ADL (Activities of Daily Living) of Katz | 6 months
  Scale measuring the autonomy of patient
Short Form 36 | 3 months
  Scale measuring the quality of life
Short Form 36 | 6 months
  Scale measuring the quality of life
Rate of patients with anterograde amnesia | 3 months
Rate of patients with anterograde amnesia | 6 months
Intracranial pressure control | 7 Days
Blood level of sodium | 7 Days
blood osmolality | 7 Days
Rate of thrombo-embolic events | 28 days
Rate of acute kidney injury | 28 days
  KDIGO 3
Rate of centropontine myelinolysis | 28 days
  Diagnosis on MRI realized in case of clinical suspicion
Blood level of chlore | 7 Days
Blood level of potassium | 5 Days
Blood level of pH (Hydrogen Potention) | 5 Days
brain oxygenation (PtiO2) | 5 Days
blood level of creatinine | 5 Days
Diuresis | 5 Days
weight | 5 Days
Ancillary study: questionnaire HADS (Hospital Anxiety and Depression Scale) in patient's relative | 6 months
  Scale measuring the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Huet, PU-PH, Principal Investigator — CHU de Brest; Lasocki Sigismond, PU-PH, Principal Investigator — University Hospital, Angers; Thomas Geerraerts, PU-PH, Principal Investigator — University Hospital, Toulouse; Francis Remerand, PU-PH, Principal Investigator — CHU de Tours; Philippe Seguin, PU-PH, Principal Investigator — Rennes University Hospital; Claire Dahyot, PU-PH, Principal Investigator — CHU Poitiers; Pierre François Perrigault, PU-PH, Principal Investigator — University Hospital, Montpellier; Jean Denis Moyer, PU-PH, Principal Investigator — AP-HP Beaujon; Tarek SHARSHAR, PU-PH, Principal Investigator — AP-HP Saint-Anne
Locations (10):
- France (10):
  - CHU Angers, Angers
  - CHU Brest Hopital La Cavale Blanche, Brest
  - AP-HP Beaujon, Clichy
  - CHU Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - Centre Hospitalier Sainte-Anne, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes-Hopital Pontchaillou, Rennes
  - CHU Toulouse Hôpital Pierre-Paul Riquet, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huet O, Chapalain X, Vermeersch V, Moyer JD, Lasocki S, Cohen B, Dahyot-Fizelier C, Chalard K, Seguin P, Hourmant Y, Asehnoune K, Roquilly A; Atlanrea Study Group and the Societe Francaise d'Anesthesie Reanimation (SFAR) Research Network. Impact of continuous hypertonic (NaCl 20%) saline solution on renal outcomes after traumatic brain injury (TBI): a post hoc analysis of the COBI trial. Crit Care. 2023 Jan 27;27(1):42. doi: 10.1186/s13054-023-04311-1. PMID 36707841
- [Derived] Roquilly A, Moyer JD, Huet O, Lasocki S, Cohen B, Dahyot-Fizelier C, Chalard K, Seguin P, Jeantrelle C, Vermeersch V, Gaillard T, Cinotti R, Demeure Dit Latte D, Mahe PJ, Vourc'h M, Martin FP, Chopin A, Lerebourg C, Flet L, Chiffoleau A, Feuillet F, Asehnoune K; Atlanrea Study Group and the Societe Francaise d'Anesthesie Reanimation (SFAR) Research Network. Effect of Continuous Infusion of Hypertonic Saline vs Standard Care on 6-Month Neurological Outcomes in Patients With Traumatic Brain Injury: The COBI Randomized Clinical Trial. JAMA. 2021 May 25;325(20):2056-2066. doi: 10.1001/jama.2021.5561. PMID 34032829
- [Derived] Roquilly A, Lasocki S, Moyer JD, Huet O, Perrigault PF, Dahyot-Fizelier C, Seguin P, Sharshar T, Geeraerts T, Remerand F, Feuillet F, Asehnoune K; COBI group. COBI (COntinuous hyperosmolar therapy for traumatic Brain-Injured patients) trial protocol: a multicentre randomised open-label trial with blinded adjudication of primary outcome. BMJ Open. 2017 Sep 24;7(9):e018035. doi: 10.1136/bmjopen-2017-018035. PMID 28947465